CLINICAL TRIAL: NCT00830388
Title: Ketoconazole Foam 2% for the Treatment of Versicolor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boni Elewski, MD (Other)
Responsible Party: Sponsor-Investigator, Boni Elewski, MD, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F080520002
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-07

CONDITIONS: Tinea Versicolor
Keywords: tinea versicolor; ketoconazole
MeSH Terms: conditions — Tinea Versicolor | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketoconazole 2% Foam (Experimental): Open-label study
  Interventions: Drug: Ketoconazole 2% Foam

INTERVENTIONS:
Drug: Ketoconazole 2% Foam — Ketoconazole 2% Foam, twice daily application to affected areas for 4 weeks.
  Other Names: Extina Foam

SUMMARY:
Ten adult patients age 19 and older with a clinical diagnosis of tinea versicolor, as well as a positive Potassium Hydroxide (KOH) using calcofluor. Ketoconazole 2% foam will be used to determine its effectiveness, safety and satisfaction when used to treat tinea versicolor.

DETAILED DESCRIPTION:
Objectives

1. To assess the efficacy of ketoconazole 2% foam for the treatment of tinea versicolor
2. To assess the safety of ketoconazole 2% foam for the treatment of tinea versicolor based on the occurrence of adverse events.
3. To assess treatment satisfaction as rated by patients

Study Design:

This will be a mono-centered, single arm, open-label pilot study. Ten adult patients age 19 and older with a clinical diagnosis of tinea versicolor, as well as a positive KOH using calcofluor, will be enrolled at the University of Alabama at Birmingham. There will be 4 scheduled visits (baseline, week 1, week 2, and week 4). A target area will be identified and mycological and clinical assessments will be performed at this site as well as a global assessment of each subject. Ketoconazole 2% foam will be applied to all affected areas for 2 weeks with a follow-up visit at week 4. Skin scraping using a disposable #15 blade for calcofluor/potassium hydroxide (KOH) assessment and photographs of target lesions will be performed at baseline, week 1, week 2, and week 4. Photographs will be taken at baseline and at week 4 (only if KOH is positive). Body surface area estimation of disease will also be performed at each visit. Evaluation of scale, hyperpigmentation/erythema, and hypopigmentation using a 4 point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) of the target area will be performed at baseline, week 1, week 2, and week 4. A global assessment will be conducted at each visit using the same 4 point scale. Patient questionnaires will be administered at baseline and week 2 to assess symptoms and satisfaction with study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 19 years and over.
2. Clinical presentation of tinea versicolor.
3. Positive KOH using calcofluor.
4. The ability to provide informed consent (including photography release)

Exclusion Criteria:

1. Use of topical antifungal to the affected area in the past 30 days
2. Use of topical steroid to the affected area in the past 14 days
3. If female, positive urine pregnancy test at screening (female patients of childbearing potential must be practicing a reliable method of birth control, not be planning a pregnancy, not be breast-feeding during the study)
4. Patients with a dermatologic condition in the region of the treatment site that in the investigator's opinion may interfere with the study results
5. Current diagnosis of immunocompromising conditions
6. Any medical or psychiatric condition that may interfere with treatment or compliance

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni E Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Dermatology, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketoconazole 2% Foam: Open-label study using Ketoconazole 2% foam applied twice daily to all affected areas for 2 weeks.
Period: Overall Study
Arm/Group | Ketoconazole 2% Foam
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketoconazole 2% Foam
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Ketoconazole 2% Foam for the Treatment of Tinea Versicolor
Description: Eleven participants were tested for the microscopic presence of yeast. At four weeks, all participants were re-tested and deemed positive if yeast continued to be present microscopically.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Ketoconazole 2% Foam
Number analyzed (Participants) | 11
participants
  Negative skin sample | 7
  Positive skin sample | 4

2. Secondary Outcome: To Assess the Safety of Ketoconazole 2% Foam for the Treatment of Tinea Versicolor Based on the Occurrence of Adverse Events.
Description: Adverse events were used to assess safety.
Time Frame: 4 weeks
Measure: Number; unit: events
Arm/Group | Ketoconazole 2% Foam
Number analyzed (Participants) | 11
events | 0

ADVERSE EVENTS:
Arm/Group | Ketoconazole 2% Foam
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes